CLINICAL TRIAL: NCT06312852
Title: Antenatal Steroids Before Elective Caesarean Section : Impact on Coagulation, Fibrinolytic System, and Other Haematological Parameters.
Brief Title: Impact of Antenatal Steroids on Coagulation.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Ahmed Mohamed Aly Ahmed Nasr, Resident of Clinical pathology department, Faculty of Medicine, Assiut University, Egypt, Assiut University
Other Study IDs: Antenatal steroids & clotting
Record Dates: First submitted 2024-03-05; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Corticosteroids Adverse Reaction
Keywords: steroid; antenatal; coagulation; fibrinolytic system; haematological parameters; hematological parameters; corticosteroid; hematological; haematological; elective; caesarean; cesarean; Fibrinolysis; Hemostasis; Plasminogen
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim of the research :

1- Detection of the presence or absence of any effect of antenatal corticosteroid administration on coagulopathy, fibrinolysis, and other haematological markers.

DETAILED DESCRIPTION:
Corticosteroid administration before anticipated preterm birth is one of the most important antenatal therapies available to improve newborn outcomes. A single course of corticosteroids is recommended for pregnant women between 28 weeks and 40 weeks of gestation who are at risk of preterm delivery within 7 days, including for those with ruptured membranes and multiple gestations (1). The administration of antenatal corticosteroids to women who, at risk of imminent preterm birth, is strongly associated with decreased neonatal morbidity and mortality (2). Neonates whose mothers received antenatal corticosteroids have significantly lower severity, frequency, or both, of respiratory distress syndrome, intracranial haemorrhage, necrotizing enterocolitis, and death, compared with neonates whose mothers did not receive antenatal corticosteroids, Betamethasone and dexamethasone are the most widely studied corticosteroids, and they generally have been preferred for antenatal treatment to accelerate foetal organ maturation (3). Both cross the placenta in their active form and have nearly identical biologic activity. Both lack mineralocorticoid activity and have relatively weak immunosuppressive activity with short-term use (4).

Increased levels of haemostatic factors, including factor VII, factor VIII, factor XI, fibrinogen, soluble CD40 ligand, and von Willebrand Factor VWF have been associated with venous and arterial thrombotic events. Similarly, impaired thrombolysis, reflected by an increase in Plasminogen activator inhibitor-1 PAI-1 levels, has been associated with adverse cardiovascular events. Although there are no previous in vivo studies in humans demonstrating that glucocorticoids directly affect haemostasis, there is in vitro and epidemiologic evidence of this phenomenon (5). In cultured human and animal cell lines, glucocorticoids increase production of von Willebrand Factor (VWF), endothelin, and PAI-1. Two studies have demonstrated dexamethasone-mediated increases in PAI-1 in cultured human adipose tissue. In patients with Cushing syndrome, elevated levels of VWF, PAI-1, thrombin-antithrombin and plasmin-antiplasmin complexes and factor VIII may resolve after curative surgical treatment. Similarly, altered levels of haemostatic factors have been reported in patients receiving exogenous glucocorticoids. The potential impact of glucocorticoids on thrombosis is clinically relevant (6). Therefore, we sought to determine the effects of antenatal glucocorticoid administration on haemostatic factors in pregnant females.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with gestational age between 28-40 weeks ( third trimester ) who will be offered antenatal steroids versus gestational-age matched controls who will not be on steroids.

Exclusion Criteria:

* Pregnant women with gestational age < 28 weeks (First trimester & Second trimester).
* Women in labour.
* Pregnant women receiving blood transfusions or on any drugs that might counteract the effect of Antenatal corticosteroids, or any drug that may have an effect on coagulation or fibrinolysis.

Ages: 15 Years to 45 Years | Sex: Female
Age Groups: Child, Adult
Study Population: Pregnant women with gestational age between 28-40 weeks ( third trimester ) who will be offered antenatal steroids ( test subjects ) versus gestational-age matched controls who will not be on steroids ( controls ).
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Antenatal corticosteroids impact on Coagulopathy | Baseline
  Detection of the presence or absence of any effect of antenatal corticosteroid administration on coagulopathy, fibrinolysis, and other haematological markers.

SECONDARY OUTCOMES:
Follow up for cases on corticosteroid therapy | Day 4
  Determine a good, feasible marker to use for follow up on cases under corticosteroid therapy.

REFERENCES:
- [Background] Obstetric Care Consensus No. 4: Periviable Birth. Obstet Gynecol. 2016 Jun;127(6):e157-e169. doi: 10.1097/AOG.0000000000001483. PMID 27214190
- [Background] Carlo WA, McDonald SA, Fanaroff AA, Vohr BR, Stoll BJ, Ehrenkranz RA, Andrews WW, Wallace D, Das A, Bell EF, Walsh MC, Laptook AR, Shankaran S, Poindexter BB, Hale EC, Newman NS, Davis AS, Schibler K, Kennedy KA, Sanchez PJ, Van Meurs KP, Goldberg RN, Watterberg KL, Faix RG, Frantz ID 3rd, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Association of antenatal corticosteroids with mortality and neurodevelopmental outcomes among infants born at 22 to 25 weeks' gestation. JAMA. 2011 Dec 7;306(21):2348-58. doi: 10.1001/jama.2011.1752. PMID 22147379
- [Background] Chawla S, Bapat R, Pappas A, Bara R, Zidan M, Natarajan G. Neurodevelopmental outcome of extremely premature infants exposed to incomplete, no or complete antenatal steroids. J Matern Fetal Neonatal Med. 2013 Oct;26(15):1542-7. doi: 10.3109/14767058.2013.791273. Epub 2013 May 7. PMID 23565886
- [Background] American College of Obstetricians and Gynecologists' Committee on Practice Bulletins-Obstetrics. Practice Bulletin No. 172: Premature Rupture of Membranes. Obstet Gynecol. 2016 Oct;128(4):e165-77. doi: 10.1097/AOG.0000000000001712. PMID 27661655
- [Background] American College of Obstetricians and Gynecologists' Committee on Practice Bulletins-Obstetrics. Practice Bulletin No. 171: Management of Preterm Labor. Obstet Gynecol. 2016 Oct;128(4):e155-64. doi: 10.1097/AOG.0000000000001711. PMID 27661654
- [Background] Kamstrup P, Rastoder E, Hellmann PH, Sivapalan P, Larsen EL, Vestbo J, Ulrik CS, Goetze JP, Knop FK, Jensen JUS. Effect of 10-Day Treatment with 50 mg Prednisolone Once-Daily on Haemostasis in Healthy Men-A Randomised Placebo-Controlled Trial. Biomedicines. 2023 Jul 21;11(7):2052. doi: 10.3390/biomedicines11072052. PMID 37509691